CLINICAL TRIAL: NCT02633670
Title: A Prospective Randomized Trial of Hemopatch Versus No Hemopatch For the Intraoperative Hemostasis During Deceased Donor Renal Transplant
Brief Title: Hemopatch Versus No Hemopatch (Renal Transplant)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Anil Kapoor, MD, FRCSC, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: TXNXHEMOPATCH
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemopatch (Experimental): The hemopatch is a promising new sealing synthetic hemostatic agent with a noval dual mechanism of action. The hemopatch is a polyethylene glycol coated (PEG coated) collagen patch. The PEG coating helps in rapid adhesion to the tissue surface while the collagen layer causes platelet activation and adhesion.
  Interventions: Device: Hemopatch
- Standard technique (Active Comparator): Standard hemostatic agents (floseal, tisseal).
  Interventions: Device: No Hemopatch

INTERVENTIONS:
Device: Hemopatch
  Arms: Hemopatch
Device: No Hemopatch
  Arms: Standard technique

SUMMARY:
Kidney transplantation remains one of the most common organ transplanted today but the surgical technique has changed very little from the original pelvic operation. The deceased donor renal transplant poses a particular challenge to the surgeon due to lack of detailed pre operative vascular assessment. The hemopatch is a promising new sealing synthetic hemostatIc agent with a novel dual mechanism of action that is more convenient to apply rather then using other hemostatic agents, which require warming and/or mixing.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age and capable of giving informed consent
* Patients scheduled for deceased donor renal transplant surgery

Exclusion Criteria:

* Patient undergoing live related transplant surgery.
* Patient having uncorrectable bleeding diathesis.
* Any patient in the no hemopatch group requiring additional haemostatic agents for achieving hemostasis like fibrillar or surgical.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Blood Loss | Baseline (Intraoperatively)
  Blood loss will be measured in ml (cc).

SECONDARY OUTCOMES:
Hemostasis achievement | Baseline (Intraoperatively)
  Hemostasis achievement will be measured in minutes.
Drop in Hemoglobin | up to 48 hours postoperatively
  Hemoglobin will be measured in g/L (drop measured from pre-operative levels to post-operative 48 hours).
Amount of Perigraft Collection | up to 48 hours postoperative
  measured in ml (with ultrasound done within 48 hours of surgery).

CONTACTS AND LOCATIONS:
Overall Officials: Anil Kapoor, MD, FRCSC, Principal Investigator — McMaster University
Locations (1):
- Marylrose Gundayao, Hamilton, Ontario, Canada